CLINICAL TRIAL: NCT02144922
Title: Effect of Pitavastatin on Coronary Flow Reserve in Hypertensive Patients With Cardiovascular Risk
Brief Title: Effect of Pitavastatin on Coronary Flow Reserve in Hypertensive Patients
Acronym: EPOCH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: JW Pharmaceutical (Industry)
Responsible Party: Principal Investigator, Duk-Hyun Kang, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013-1091
Record Dates: First submitted 2014-05-20; First posted 2014-05-22 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Hypertension; Cardiovascular Risk
Keywords: Hypertension; Statin
MeSH Terms: conditions — Hypertension | interventions — pitavastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): Patients continue taking their antihypertensive medication alone.
  Interventions: Other: Control
- Pitavastatin (Active Comparator): Pitavastatin 4 mg is given to study patients after a baseline assessment and continued for 1 year without further dose titration. Patients continue taking their antihypertensive medication during the entire follow-up period.
  Interventions: Drug: Pitavastatin

INTERVENTIONS:
Drug: Pitavastatin — statin
  Other Names: Livalo
  Arms: Pitavastatin
Other: Control — Life style modification alone
  Arms: Control

SUMMARY:
Although statins reduce cardiac events in hypertensive patients with cardiovascular risk factors, the effect of statins on coronary flow reserve (CFR) has not been examined in such patients. The investigators hypothesize that pitavastatin added to standard antihypertensive therapy will be superior to placebo in improving CFR in hypertensive patients with cardiovascular risk, and try to examine this hypothesis in a double-blind, randomized comparison study using Doppler echocardiography.

DETAILED DESCRIPTION:
Statin treatment improves coronary flow reserve (CFR) and decreases cardiac morbidity and mortality in patients with coronary artery disease (CAD) and hypercholesterolemia. Endothelial dysfunction and impairment in coronary microcirculation is also observed in hypertensive patients with cardiovascular risk factors. However, the measurement of CFR has rarely been performed in hypertensive patients without CAD, because CFR could be invasively measured using a Doppler guide wire in a cardiac catheterization laboratory. Recent advances in echocardiographic imaging techniques have made it possible to measure coronary flow velocity and CFR, which highly correlates with the CFR measured by invasive means.

Lipid lowering with a statin provided beneficial effects in patients with average levels of serum total cholesterol in the Anglo-Scandinavian Cardiac Outcomes Trial-Lipid Lowering Arm (ASCOT-LLA) study conducted in hypertensive patients at cardiovascular risk. Improvements in endothelial dysfunction and CFR may be related to the beneficial effects of statins in hypertensive patients without hypercholesterolemia, but the effect of statins on CFR has not been examined in such patients. Accordingly, the investigators try to examine the hypothesis that pitavastatin added to standard antihypertensive therapy in hypertensive patients with cardiovascular risk will be superior to placebo in improving CFR in a double-blind, randomized comparison study using Doppler echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* Controlled Hypertension: treated SBP<140 mmHg and DBP<90 mmHg
* LDL cholesterol ≥ 130mg/dL
* Patients with statin-naive state, defined as receiving no statin therapy for more than 6 months during the previous 12 months.
* Any 1 of these cardiovascular risk factors required: smoking, age over 55 (men) or 65 (women), history of cerebrovascular event, family history of early CHD before age 55, HDL cholesterol < 40 mg/dL

Exclusion Criteria:

* A previous history of intolerance or hypersensitivity to statins
* Uncontrolled hypertension; SBP≥140 mmHg or DBP≥90 mmHg
* Previous MI or currently treated angina pectoris
* Stroke, TIA < 3 months
* Secondary hypertension
* Fasting serum triglyceride > 500 mg/dL
* Clinical congestive heart failure
* Uncontrolled arrhythmia
* Left ventricular hypertrophy: LV mass index >134g/m2 (male) or >110g/m2 (female)
* Concomitant clinically important hematological, gastrointestinal, hepatic, renal or other disease
* Pregnant or lactating women and those of child-bearing potential
* Diabetes
* Peripheral vascular disease
* Unwillingness or inability to comply with the procedures described in this protocol

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2014-05; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
change in the CFR value | 12 months
  Change of coronary flow velocity reserve from baseline to 1 year follow-up. For each patient, the averaged value of coronary flow velocity reserve will be obtained at baseline and 1 year follow-up.
Difference in mean CFR value | 12 months
  DIfference in CFR value at 12 month follow-up between pitavastatin and placebo arm

SECONDARY OUTCOMES:
change of CRP | 12 months
  Change of CRP from baseline to 1 year follow-up.
Change of LDL-cholesterol | 12 months
  Change of LDL-cholesterol from baseline to 1 year follow-up.
Change of averaged peak diastolic velocity | 12 months
  Change of averaged peak diastolic velocity from baseline to study end.

CONTACTS AND LOCATIONS:
Overall Officials: Duk-Hyun Kang, M.D., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No